CLINICAL TRIAL: NCT06918561
Title: A Randomized Controlled Multisite Crossover Trial Evaluating the Efficacy of NeoThelium FT in the Treatment of "Other" Open Wounds
Brief Title: Evaluating the Efficacy of NeoThelium FT in the Treatment of Chronic Open Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NuScience Medical Biologics, LLC (Industry)
Collaborators: SygNola, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HEAL
Record Dates: First submitted 2025-03-31; First posted 2025-04-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Open Wound
Keywords: Chronic wounds; Wound Medicine; Cellular, Acellular, Matrix-like Product (CAMP); Cellular and/or Tissue Product (CTP); Dehydrated Complete Human Placental Membrane (dCHPM)
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The subject will be randomized to one of the following treatments:
  * Standard of care
  * NeoThelium FT in addition to standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Standard of Care (Active Comparator): Wound cleansing, Sharps debridement, Dressing for moisture balance, Offloading
  Interventions: Other: Standard of Care
- Intervention: NeoThelium FT & Standard of Care (Experimental): Wound cleansing, sharps debridement, NeoThelium FT application, Dressing for moisture balance, Offloading
  Interventions: Other: NeoThelium FT

INTERVENTIONS:
Other: Standard of Care — Wound cleansing, Sharps debridement, Dressing for moisture balance, Offloading
  Arms: No Intervention: Standard of Care
Other: NeoThelium FT — NeoThelium FT is a dehydrated wound covering derived from donated human placental tissue. NeoThelium FT is a dual-layer membrane with amnion and chorion combination layers.
  Arms: Intervention: NeoThelium FT & Standard of Care

SUMMARY:
This is a randomized controlled crossover trial evaluating the efficacy of NeoThelium FT in conjunction with standard of care vs. standard of care alone in treating chronic open wounds.

DETAILED DESCRIPTION:
This research will take place across multiple medical centers, where both researchers and participants will know which treatment is being used (open label). Patients who agree to participate and meet the study requirements during screening will be randomly assigned to one of two groups: either standard of care (SOC) alone, or SOC plus NeoThelium FT.

The study includes a crossover component for subjects in the SOC arm. At treatment visit 13 (approximately 84 days post-randomization), SOC arm subjects not having achieved complete wound closure, and still meeting the inclusion/exclusion criteria, are eligible to cross over to the IP arm (SOC plus NeoThelium FT). Crossover subjects will begin IP arm treatment with weekly NeoThelium FT applications for up to 12 treatment visits. The subject will continue follow-up per the original schedule. As this is a post-marketing study, it will gather information regarding the efficacy of treatment while also supporting insurance reimbursement decisions. All subjects will complete two-week screening phase prior to being randomized into a treatment arm. Treatment arms will consist of NeoThelium FT in conjunction with standard of care, vs. standard of care alone. The primary endpoint will be the percentage of target ulcers that achieve complete wound closure within 12 weeks. Secondary endpoints consist of wound percentage area reduction rates and pain assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 years of age or older
2. Subject has a medical diagnosis of "other" Open wound
3. Subject has a chronic open wound present for 4 weeks or greater (documented in medical record), and less than 12 months duration if being treated with continuous SOC
4. Subject has a chronic open wound with a historical wound measurement showing less than 25% healing within 14 days prior to screening
5. Subject has a chronic open wound with screening wound measurement showing less than 25% healing within 14 days prior to randomization
6. Subject has an Open wound without infection or clinically visible exposed bone
7. Index wound is a minimum of 0.5cm2 and a maximum of 25cm2 at first treatment visit
8. Index ulcer has a maximum depth of 1cm at screening visit 1
9. The chronic open wound is treated with offloading therapy, if applicable to location, while standing, sitting, and lying down for 14 days prior to randomization
10. Adequate circulation of wounds located below the knee demonstrated by an ABI of >0.7 and <1.3, or TBI of >0.6 within 30 days prior to randomization OR an arterial ultrasound noted with patent circulation and without significant stenosis 90 days prior to randomization.
11. Index ulcer is free of infection prior to randomization and during screening phase.
12. Index ulcer is free of necrotic debris prior to NeoThelium FT application
13. Female subjects of childbearing potential having a negative pregnancy test prior to randomization
14. Index ulcer is free of infection prior to randomization and during screening phase noted with the NERDS Assessment. Infection must be adequately treated and controlled prior to randomization.
15. Subject is able and willing to follow the protocol requirements
16. Subject had signed informed consent
17. If 2 or more ulcers are present, the ulcers must be separated by at least 2 cm

Exclusion Criteria:

1. Subject with a wound diagnosis of diabetic foot wound, pressure wound, venous leg wound, burn wound, or alternative diagnosis other than "open wound"
2. Subject has a known life expectancy of <1 year
3. Subject is unable to comply with protocol treatment
4. Subject has major uncontrolled medical disorders in the opinion of the investigator, such as serious cardiovascular, renal, liver, pulmonary, autoimmune, palliative care, or inherited blood disorders that may affect wound healing.
5. Subject actively being treated for malignant disease or history of malignancy or radiation therapy at the site of wound
6. Subject has comorbid conditions that may compromise subject safety in the opinion of the investigator
7. Known contraindications to tissue-engineered allograft
8. Concurrent participation in alternative clinical trial that involves investigational drug or product interfering with wound treatment and/or healing
9. Subject is pregnant or breastfeeding
10. Subject with history of immunosuppressant treatment (systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or topical steroid application to the wound surface for >2 weeks duration within 30 days prior to randomization; or anticipated use of the above during the course of the study
11. Wound previously treated with CAMPs, tissue engineered, or scaffold materials within 30 days prior to randomization
12. Open wound with active infection
13. Wound depth with visible exposed bone
14. HBOT within 14 days prior to randomization
15. Revascularization surgery on the index wound leg within 30 days of screening phase
16. Index wound suspicious of neoplasm in the opinion of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Complete Wound Closure | 1-12 weeks
  The primary endpoint will be the percentage of target ulcers that achieve complete wound closure.

SECONDARY OUTCOMES:
Percentage Wound Area Change | 1-12 weeks
  The percentage change in wound area from TV-1 to TV-13 will be measured weekly using digital photographic planimetry and physical examination.
Pain Assessment | Day 0, Day 14, Day 35, Day 56, Day 84
  Change in pain associated with the target ulcer will be assessed using the Numeric Pain Rating Scale at designated time points

OTHER OUTCOMES:
Adverse Events and Serious Adverse Events | Day -14 through 91 days
  The number and nature of adverse events (AEs) and series adverse events (SAEs) occurring during the study will be tracked and reported.
Follow-Up Closure | 2 weeks
  Number of wounds remaining closed during the 2-week follow-up
Time to Closure | 1-12 weeks
  Average number of grafts and/or weeks used to achieve wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Angelina Ferguson, DNP, Study Director — SygNola, LLC
Locations (3):
- United States (3):
  - MedCentris of Hammond, Hammond, Louisiana
  - MedCentris of Slidell, Slidell, Louisiana
  - MedCentris of D'iberville, D'Iberville, Mississippi

IPD SHARING:
Plan to Share IPD: No